CLINICAL TRIAL: NCT02940704
Title: Assessment of Postoperative Pain After Using Reciproc Versus One Shape NiTi Systems in Patients With Symptomatic Irreversible Pulpitis: A Randomized Clinical Trial (Part I)
Brief Title: Assessment of Postoperative Pain After Using Reciproc Versus One Shape NiTi Systems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Michel Karam Eissa Elias, Resident at endodontic department - Faculty of Oral and Dental Medicine- Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEBC-CU-2016-10-145
Record Dates: First submitted 2016-10-18; First posted 2016-10-21 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Pulpitis
Keywords: Reciproc; One Shape; reciprocation; continuous rotation; irreversible pulpitis; postoperative pain
MeSH Terms: conditions — Pulpitis; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Reciproc (Experimental): * Reciproc (VDW, Munich, Germany) is a single file reciprocating system for mechanical instrumentation of root canals.
  * Size: R40 (40/0.06)
  Interventions: Procedure: Reciproc
- One Shape (Active Comparator): * One Shape (MicroMega, Besançon Cedex, France) is a single file system that works by continuous rotation for mechanical instrumentation of root canals.
  * Size: 25/0.06
  Interventions: Procedure: One Shape

INTERVENTIONS:
Procedure: Reciproc — * Canals will be instrumented using Reciproc reciprocating system set on an electric motor, with adjusted torque and speed according to the manufacturer's instructions.
  * There is no need for coronal preflaring with a Gates Glidden drill or an orifice opener since the design of the Reciproc instrument allows any obstructions in the coronal third to be removed, as claimed by the manufacturer.
  * Reciproc file selection: R40 (40/0.06) is to be used.
  Arms: Reciproc
Procedure: One Shape — * Coronal preflaring will be performed using Gates Glidden drill.
  * Canals will be instrumented using One Shape single-file (25/0.06) set on an electric motor with adjusted torque and speed according to the manufacturer's instructions.
  * For wide canals, One Shape Apical (30/0.06, 37/0.06) will be used.
  Arms: One Shape

SUMMARY:
* The aim of this study is to assess the postoperative pain and the intake of analgesic medication after using Reciproc single-file reciprocating system or One Shape single-file continuous rotary system in patients with symptomatic irreversible pulpitis.
* Patients will be diagnosed to determine whether they are eligible for the inclusion criteria of this study or not. Patients who are eligible will then start their root canal treatment on the same visit and to be completed in one visit only. Patients will be phone called in order to record the intensity of pain, amount and frequency of analgesic intake at 6, 12, 24, 48 and 72 hours after treatment.

DETAILED DESCRIPTION:
- Full medical and dental history using a schematic dental chart will be obtained from all eligible participants. Each tooth will be evaluated for vitality (sensitivity) of pulp tissues.

The patients will be randomly divided into 2 groups:

* Experimental group: Reciproc reciprocating instrumentation system.
* Control group: One Shape rotary instrumentation system.

  - Sequence of Procedural steps
  1. Preoperative pain will be assessed by Numerical Rating Scale (NRS) before administration of anesthesia.
  2. Local anesthesia will be achieved using 2% lidocaine (1:100,000 adrenaline).
  3. An access cavity will be performed using round bur and Endo-Z bur.
  4. The tooth will be properly isolated with rubber dam.
  5. Working length will be determined using an electronic apex locator, and working length will be confirmed by radiograph using K-file. Then the working length will be established at 0.5 mm up to the radiographic apex.
  6. Canals will be explored with hand K-file ISO sizes 10, 15, 20.
  7. Mechanical preparation for both groups will be as follows:
* Experimental group:

  * Canals will be instrumented using Reciproc reciprocating system set on an electric motor, with adjusted torque and speed according to the manufacturer's instructions.
  * There is no need for coronal preflaring with a Gates Glidden drill or an orifice opener since the design of the Reciproc instrument allows any obstructions in the coronal third to be removed, as claimed by the manufacturer.
  * Reciproc file selection: R40 (40/0.06) is to be used.
* Control group:

  * Coronal preflaring will be performed using Gates Glidden drill.
  * Canals will be instrumented using One Shape (25/0.06) set on an electric motor with adjusted torque and speed according to the manufacturer's instructions.
  * For wide canals, One Shape Apical (30/0.06, 37/0.06) will be used.

    8.The rotary files will be introduced inside the canal using EDTA gel. 9.Canals will be irrigated with 2.5% sodium hypochlorite solution between every subsequent instrument. It is prepared by adding 10 ml of sterile distilled water to 10 ml of 5.25% sodium hypochlorite solution using a 27-gauge needle fit to 5 ml disposable plastic syringe placed as far as possible in the canal space without binding.

    10.Canals will be dried with sterile paper points and obturated using lateral condensation technique. A spreader will be used to allow space for auxiliary cones, with resin-based root canal sealer.

    11.The tooth will be sealed by temporary restoration, and postoperative pain will be assessed immediately after the end of treatment.

    12.The patient will be instructed to return to complete the treatment procedures until placing a full-coverage restoration.

    13.The patient will be instructed to take one tablet 400 mg Ibuprofen if he/she experiences severe pain.

ELIGIBILITY:
Inclusion Criteria:

Single-rooted mandibular premolar teeth with:

* Preoperative sharp pain.
* Vital response of pulp tissue.
* Normal periapical radiographic appearance or slight widening in lamina dura.

Exclusion Criteria:

i. Patients who have already consumed preoperative medication, such as analgesic, non-steroidal or steroidal anti-inflammatory drugs, within 12 hours before treatment.

ii. Patients who have more than one tooth in the same quadrant and/or opposite quadrant that require an endodontic treatment.

iii. Pregnant females. iv. Patients having significant systemic disorder. v. If antibiotics have been administrated during the past two weeks preoperatively.

vi. Patients having bruxism or clenching. vii. Teeth that have:

* Non vital pulp tissues.
* Association with swelling or fistulous tract.
* Pocket depth greater than 5 mm.
* Previous endodontic treatment.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
postoperative pain | Up to 72 hrs after treatment
  Intensity of pain after endodontic treatment by Numerical Rating Scale (0-10)

SECONDARY OUTCOMES:
Number of analgesic tablets taken after endodontic treatment | up to 72 hours after treatment
  One tablet 400 mg Ibuprofen if patient experiences severe pain after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Michel K Elias, Resident, Principal Investigator — Faculty of Oral and Dental Medicine - Cairo University; Hebatallah M El-Far, Professor, Study Director — Faculty of Oral and Dental Medicine - Cairo University; Shaimaa I Gawdat, Lecturer, Study Chair — Faculty of Oral and Dental Medicine - Cairo University
Locations (1):
- Endodontic Department - Faculty of Oral and Dental Medicine - Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shahi S, Asghari V, Rahimi S, Lotfi M, Samiei M, Yavari H, Shakouie S, Nezafati S. Postoperative Pain after Endodontic Treatment of Asymptomatic Teeth Using Rotary Instruments: A Randomized Clinical Trial. Iran Endod J. 2016 Winter;11(1):38-43. doi: 10.7508/iej.2016.01.008. Epub 2015 Dec 24. PMID 26843876
- [Background] Shokraneh A, Ajami M, Farhadi N, Hosseini M, Rohani B. Postoperative endodontic pain of three different instrumentation techniques in asymptomatic necrotic mandibular molars with periapical lesion: a prospective, randomized, double-blind clinical trial. Clin Oral Investig. 2017 Jan;21(1):413-418. doi: 10.1007/s00784-016-1807-2. Epub 2016 Apr 4. PMID 27041109
- [Background] Caviedes-Bucheli J, Azuero-Holguin MM, Gutierrez-Sanchez L, Higuerey-Bermudez F, Pereira-Nava V, Lombana N, Munoz HR. The effect of three different rotary instrumentation systems on substance P and calcitonin gene-related peptide expression in human periodontal ligament. J Endod. 2010 Dec;36(12):1938-42. doi: 10.1016/j.joen.2010.08.043. Epub 2010 Oct 15. PMID 21092809
- [Background] Haapasalo, M. & Shen, Y. Evolution of nickel-titanium instruments: from past to future. Endod. Top. 29, 3-17 (2013).
- [Background] Kucukyilmaz E, Savas S, Saygili G, Uysal B. Assessment of apically extruded debris and irrigant produced by different nickel-titanium instrument systems. Braz Oral Res. 2015;29:1-6. doi: 10.1590/1807-3107bor-2015.vol29.0002. Epub 2014 Nov 11. PMID 25387860
- [Background] Kherlakian D, Cunha RS, Ehrhardt IC, Zuolo ML, Kishen A, da Silveira Bueno CE. Comparison of the Incidence of Postoperative Pain after Using 2 Reciprocating Systems and a Continuous Rotary System: A Prospective Randomized Clinical Trial. J Endod. 2016 Feb;42(2):171-6. doi: 10.1016/j.joen.2015.10.011. Epub 2015 Nov 29. PMID 26614017
- [Background] Gambarini, D. G. & Glassman, G. Continuing education TF Adaptive : a novel approach to nickel-titanium instrumentation. Oral Heal. J. (2013).
- [Background] Nekoofar MH, Sheykhrezae MS, Meraji N, Jamee A, Shirvani A, Jamee J, Dummer PM. Comparison of the effect of root canal preparation by using WaveOne and ProTaper on postoperative pain: a randomized clinical trial. J Endod. 2015 May;41(5):575-8. doi: 10.1016/j.joen.2014.12.026. Epub 2015 Feb 24. PMID 25720984
- [Background] Gambarini G, Testarelli L, De Luca M, Milana V, Plotino G, Grande NM, Rubini AG, Al Sudani D, Sannino G. The influence of three different instrumentation techniques on the incidence of postoperative pain after endodontic treatment. Ann Stomatol (Roma). 2013 Mar 20;4(1):152-5. doi: 10.11138/ads.0152. Print 2013 Jan. PMID 23741536
- [Background] Neelakantan P, Sharma S. Pain after single-visit root canal treatment with two single-file systems based on different kinematics--a prospective randomized multicenter clinical study. Clin Oral Investig. 2015 Dec;19(9):2211-7. doi: 10.1007/s00784-015-1448-x. Epub 2015 Mar 15. PMID 25773449
- [Background] Relvas JB, Bastos MM, Marques AA, Garrido AD, Sponchiado EC Jr. Assessment of postoperative pain after reciprocating or rotary NiTi instrumentation of root canals: a randomized, controlled clinical trial. Clin Oral Investig. 2016 Nov;20(8):1987-1993. doi: 10.1007/s00784-015-1692-0. Epub 2015 Dec 19. PMID 26685850